CLINICAL TRIAL: NCT01394289
Title: Biological Standardization of Lolium Perenne Allergen Extract to Determine the Biological Activity in HEP Units
Brief Title: Biological Standardization of Lolium Perenne Allergen Extract
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Laboratorios Leti, S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 6041-PR-PRI-182; 2010-023949-29
Record Dates: First submitted 2011-07-13; First posted 2011-07-14 (Estimated); Last update posted 2012-08-27 (Estimated); Status verified 2011-08

CONDITIONS: Allergy to Grass Pollen
Keywords: Standardization; Immunotherapy; Skin prick test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Biological/Vaccine: Lolium allergen extract (Experimental): Four concentrations of Lolium perenne allergen extract, together with a positive and negative control, using 10 mg/ml histamine dihydrochloride solution and a glycerinated phenol saline solution, respectively, will be tested in every patient in duplicate on the volar surface of the forearm. This test will be referred to as the Titrated Skin Prick test.
  Interventions: Biological: Lolium allergen extract

INTERVENTIONS:
Biological: Lolium allergen extract — This is an open, unblinded and non randomized biological as proposed by the Nordic Guidelines.
  Four concentrations of Lolium perenne allergen extract, together with a positive and negative control, using 10 mg/ml histamine dihydrochloride solution and a glycerinated phenol saline solution, respectively, will be tested in every patient in duplicate on the volar surface of the forearm. This test will be referred to as the Titrated Skin Prick test.

SUMMARY:
The objective of this study is to determine the biologic activity of a Lolium perenne allergen extract in histamine equivalent prick (HEP) units, in order to be used as in-house reference preparation (IHRP).

DETAILED DESCRIPTION:
Four concentrations of Lolium perenne allergen extract, together with a positive and negative control, using 10 mg/ml histamine dihydrochloride solution and a glycerinated phenol saline solution, respectively, will be tested in every patient in duplicate on the volar surface of the forearm.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided written informed consent, appropriately signed and dated by the subject (or legal representative, if applicable).
* Subject can be male or female of any race and ethnic group.
* Age > 18 years and < 50 years at the study inclusion day.
* Positive skin prick test with a standardized commercially available preparation of Lolium perenne allergen extract. The skin prick test will be considered positive if the test results in a wheal major diameter of at least 3 mm and at least the size of the positive control. Positive skin prick test results are valid if performed within one year prior to the inclusion of the subject in the study
* A positive test for specific IgE to Lolium perenne (CAP-RAST ≥ 2). IgE results are valid if performed within one year prior to the inclusion of the subject in the study.
* Allergic symptoms during the pollen season of Lolium perenne.
* Mean of the forearm major diameters of the wheals provoked by histamine dihydrochloride (10 mg/ml) ≥ 3 mm.

Exclusion Criteria:

* Immunotherapy in the past 5 years with an allergen preparation known to interfere with the allergen to be tested (e.g., grass group extracts).
* Use of drugs that may interfere with the skin reactions (e.g., antihistamines). See Appendix 1
* Treatment with any of the following medications: tricyclic or tetracyclic antidepressants, β-blockers or corticosteroids (> 10 mg/day of prednisone or equivalent).
* Pregnancy.
* Dermographism affecting the skin area at the test site at either study visit.
* Atopic dermatitis affecting the skin area at the test site at either study visit.
* Urticaria affecting the skin area at the test site at either study visit.
* Participation in another clinical trial within the last month.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2011-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Wheal size area (mm2) on the skin at the site of the puncture during the immediate phase. | 30 minutes per subject

CONTACTS AND LOCATIONS:
Overall Officials: María José Gómez, Study Chair — Laboratorios LETI, S.L.U
Locations (2):
- Spain (2):
  - Hospital Universitario de Salamanca, Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocío, Seville, Sevilla